CLINICAL TRIAL: NCT04074317
Title: A Phase 2, Single-Dose, Randomized, Open-Label, Active-Controlled, Crossover, Pharmacodynamic, and Pharmacokinetic Comparative Study of a Novel Pramlintide-Insulin Co-Formulation in Adults With Type 1 Diabetes Mellitus
Brief Title: Phase 2, Randomized, Open-Label, Crossover, PD/PK Study of a Novel Pram-Insulin Co-Formulation in Adults With T1D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DPI-201
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1; Insulin-dependent Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin; pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- PRAM9 to Regular Insulin to Regular Insulin+pramlintide (Experimental): Xeris pramlintide + insulin co-formulation (PRAM9) to Regular Insulin (Humulin®) to Regular Insulin+pramlintide (Symlin® pen) as separate SC injections
  Interventions: Drug: PRAM9; Drug: Regular Insulin + Pramlintide; Drug: Regular Insulin
- Regular Insulin to Regular Insulin+pramlintide to PRAM9 (Experimental): Regular Insulin (Humulin®) to Regular Insulin+pamlintide (Symlin® pen) as separate SC injections to PRAM9
  Interventions: Drug: PRAM9; Drug: Regular Insulin + Pramlintide; Drug: Regular Insulin
- Regular Insulin+pramlintide to PRAM9 to Regular Insulin (Experimental): Regular Insulin (Humulin®)+pramlintide (Symlin® pen) as separate SC injections to Xeris pramlintide + insulin co-formulation (PRAM9) to Regular Insulin
  Interventions: Drug: PRAM9; Drug: Regular Insulin + Pramlintide; Drug: Regular Insulin
- PRAM9 to Regular Insulin+pramlintide to Regular Insulin (Experimental): Xeris pramlintide + insulin co-formulation (PRAM9) to Regular Insulin (Humulin®)+pramlintide (Symlin® pen) as separate SC injections to Regular Insulin
  Interventions: Drug: PRAM9; Drug: Regular Insulin + Pramlintide; Drug: Regular Insulin
- Regular Insulin to PRAM9 to Regular Insulin+pramlintide (Experimental): Regular Insulin (Humulin®) to Xeris pramlintide + insulin co-formulation (PRAM9) to Regular Insulin+pramlintide (Symlin® pen) as separate SC injections to Regular Insulin
  Interventions: Drug: PRAM9; Drug: Regular Insulin + Pramlintide; Drug: Regular Insulin
- Regular Insulin+pramlintide to Regular Insulin to PRAM9 (Experimental): Regular Insulin (Humulin®)+pramlintide (Symlin® pen) as separate SC injections to Xeris pramlintide + insulin co-formulation (PRAM9) to Regular Insulin to Xeris pramlintide + insulin co-formulation (PRAM9)
  Interventions: Drug: PRAM9; Drug: Regular Insulin + Pramlintide; Drug: Regular Insulin

INTERVENTIONS:
Drug: PRAM9 — SC injection
Drug: Regular Insulin + Pramlintide — Separate SC injections
Drug: Regular Insulin — SC injection

SUMMARY:
This is a randomized, open-label, active-controlled, single-dose, 3-treatment, 3-period, 3-way crossover, comparative PD and PK inpatient study in adults with T1D. The study comprises 5 visits: Screening (Visit 1), Treatment Periods (Visits 2 - 4), and Follow-Up (Visit 5).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the PD properties of a single dose of PRAM9 compared to single doses of regular insulin and regular insulin plus pramlintide (co-administered as separate injections) in adults with T1D. The secondary objectives of this study are to evaluate the safety and PK profiles of a single dose of PRAM9 compared to single doses of regular insulin and regular insulin plus pramlintide (co-administered as separate injections) in adults with T1D. During each treatment period subjects will receive a single SC dose of PRAM9, regular insulin, or co-administered regular insulin plus pramlintide.

ELIGIBILITY:
Inclusion Criteria:

1. Understands the study procedures, alternative treatment available, and risks involved with the study, and voluntarily agrees to participate by giving written informed consent
2. Male or non-pregnant, non-lactating female diagnosed with T1D for at least 24 months prior to Screening.
3. Aged 18 to 64 years of age, inclusive
4. On a stable insulin regimen for 21 days prior to Screening (no greater than ± 20% variability in total daily dose)
5. Have a plasma C-peptide level < 0.6 ng/mL at Screening
6. Have an HbA1c < 10% at Screening
7. Body mass index (BMI) in the range of ≥ 18 to ≤ 35 kg/m2 at Screening
8. For women of childbearing potential, there is a requirement for a negative urine pregnancy test at Screening and for agreement to use contraception throughout the study and for 7 days after the last dose of study drug. Acceptable contraception includes birth control pill/patch/vaginal ring, Depo-Provera® (medroxyprogesterone acetate), Norplant® System (levonorgestrel), an intra-uterine device (IUD), the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
9. Fasting Serum triglyceride concentration < 200 mg/dL

Exclusion Criteria:

1. Currently being treated with pramlintide or has discontinued pramlintide within 21 days of Screening
2. Currently using an insulin pump
3. Has renal insufficiency (serum creatinine <3.0 mg/dL) or end-stage renal disease requiring renal replacement therapy
4. Has hepatic disease, including serum ALT or AST ≥3 times the upper limit of normal (ULN)
5. Has hepatic synthetic insufficiency (serum albumin <3.0 g/dL)
6. Has a hematocrit value that is exclusionary: Female <35.5% and Male <38.3%
7. Has a hemoglobin value that is exclusionary: Female <11.5 g/dL and Male <12.5 g/dL
8. Has out-of-range systolic or diastolic BP readings at Screening (systolic BP <90 or >150 mm Hg or diastolic BP <50 or >100 mm Hg)
9. Has clinically significant ECG abnormalities at Screening
10. Has congestive heart failure, NYHA Class III or IV
11. Has history of myocardial infarction, unstable angina, or revascularization within 6 months prior to Screening
12. Has history of a cerebrovascular accident in 6 months prior to Screening with major neurological deficits
13. Has active malignancy within 5 years prior to Screening (exception: basal cell or squamous cell skin cancers)
14. Has had major surgical operation within 60 days prior to Screening or planned surgical operation during the study
15. Has a seizure disorder (other than with suspected or documented hypoglycemia)
16. Has a current bleeding disorder, treatment with anticoagulants, or platelet count <50 ×10^9/L
17. Has a history of allergies or significant hypersensitivity to pramlintide or any pramlintide-related products or to any of the excipients in the investigational formulation
18. Has a history of positive test result for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
19. Has a concurrent illness not controlled by a stable therapeutic regimen
20. Tests positive for drugs of abuse at Screening. Subjects testing positive for tetrahydrocannabinol (THC) at Screening or reporting active marijuana use will be allowed to participate in the study at the discretion of the investigator.
21. Has active substance or alcohol abuse (>21 drinks/week for males or >14 drinks/week for females)
22. Has participated in other studies involving administration of an investigational drug within 30 days or 5 half-lives prior to Screening (whichever is longer) or during participation in the current study
23. There is any reason the investigator deems exclusionary
24. Has donated blood within 8 weeks prior to Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Valasquez, Study Director — Worldwide Clinical Trials; George Atiee, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- World Wide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a 3-treatment, 6-sequence, 3-period crossover design where 18 eligible subjects randomized to 6 treatment sequences (3 subjects per sequence), with each subject scheduled to receive all 3 treatments.
Groups:
- PRAM9 to Regular Insulin to Regular Insulin+Pramlintide; Regular Insulin to Regular Insulin+Pramlintide to PRAM9; Regular Insulin+Pramlintide to PRAM9 to Regular Insulin; PRAM9 to Regular Insulin+Pramlintide to Regular Insulin; Regular Insulin to PRAM9 to Regular Insulin+Pramlintide; Regular Insulin+Pramlintide to Regular Insulin to PRAM9: PRAM9 (Xeris pramlintide + insulin co-formulation): SC injection Regular Insulin (Humulin®): SC injection Regular Insulin (Humulin®) + Pramlintide (Symlin®): Separate SC injections
Period: First Period
Arm/Group | PRAM9 to Regular Insulin to Regular Insulin+Pramlintide | Regular Insulin to Regular Insulin+Pramlintide to PRAM9 | Regular Insulin+Pramlintide to PRAM9 to Regular Insulin | PRAM9 to Regular Insulin+Pramlintide to Regular Insulin | Regular Insulin to PRAM9 to Regular Insulin+Pramlintide | Regular Insulin+Pramlintide to Regular Insulin to PRAM9
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Period
Arm/Group | PRAM9 to Regular Insulin to Regular Insulin+Pramlintide | Regular Insulin to Regular Insulin+Pramlintide to PRAM9 | Regular Insulin+Pramlintide to PRAM9 to Regular Insulin | PRAM9 to Regular Insulin+Pramlintide to Regular Insulin | Regular Insulin to PRAM9 to Regular Insulin+Pramlintide | Regular Insulin+Pramlintide to Regular Insulin to PRAM9
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Period
Arm/Group | PRAM9 to Regular Insulin to Regular Insulin+Pramlintide | Regular Insulin to Regular Insulin+Pramlintide to PRAM9 | Regular Insulin+Pramlintide to PRAM9 to Regular Insulin | PRAM9 to Regular Insulin+Pramlintide to Regular Insulin | Regular Insulin to PRAM9 to Regular Insulin+Pramlintide | Regular Insulin+Pramlintide to Regular Insulin to PRAM9
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics by enrollment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRAM9 to Regular Insulin to Regular Insulin+Pramlintide | Regular Insulin to Regular Insulin+Pramlintide to PRAM9 | Regular Insulin+Pramlintide to PRAM9 to Regular Insulin | PRAM9 to Regular Insulin+Pramlintide to Regular Insulin | Regular Insulin to PRAM9 to Regular Insulin+Pramlintide | Regular Insulin+Pramlintide to Regular Insulin to PRAM9 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 3 | 3 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (21.36) | 45.0 (18.68) | 42.3 (14.50) | 38.0 (5.57) | 42.0 (9.54) | 49.3 (4.73) | 43.9 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 3 | 2 | 1 | 10
  Male | 3 | 1 | 1 | 0 | 1 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 2 | 1 | 6
  Not Hispanic or Latino | 3 | 3 | 2 | 1 | 1 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 2 | 3 | 3 | 3 | 3 | 3 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 18
Weight [Mean (Standard Deviation); unit: kg] | 81.30 (4.952) | 72.23 (2.902) | 83.43 (22.74) | 62.27 (4.099) | 76.20 (11.888) | 80.53 (11.869) | 75.99 (12.407)
Height [Mean (Standard Deviation); unit: cm] | 175.43 (7.643) | 173.20 (15.552) | 170.47 (14.332) | 160.17 (5.299) | 169.17 (17.208) | 175.00 (9.034) | 170.57 (11.642)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.543 (3.060) | 24.340 (3.196) | 28.267 (3.248) | 24.313 (2.039) | 26.620 (1.257) | 26.183 (1.669) | 26.044 (2.562)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0-180 Minutes for Plasma Glucose >180 mg/dL
Description: The PD effects on plasma glucose levels were compared among the treatment arms as defined by AUC0-180 (mg/dL * minutes) for plasma glucose >180 mg/dL
Time Frame: 0-180 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants with glucose >180 mg/dL.
Measure: Mean (Standard Deviation); unit: min*mg/dL
Groups:
- PRAM9: PRAM9 (Xeris pramlintide + insulin co-formulation): SC injection
- Regular Insulin + Pramlintide: Regular Insulin (Humulin®) + Pramlintide (Symlin®): Separate SC injections
- Regular Insulin: Regular Insulin (Humulin®): SC injection
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 14 | 16 | 14
min*mg/dL | 5019.6 (4276.53) | 4591.9 (3095.53) | 13317.5 (5262.42)
Statistical Analysis 1: Comparison: PRAM9 vs Regular Insulin; Test type: Equivalence — Treatment groups were compared using an analysis of variance (ANOVA) model, including sequence, period, and treatment as fixed effects and patient within sequence as random effect; p < 0.0001, ANOVA — Least-squares geometric means for ln-transformed data
Statistical Analysis 2: Comparison: PRAM9 vs Regular Insulin + Pramlintide; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.694, ANOVA
Statistical Analysis 3: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA

2. Secondary Outcome: Mean Proportional Time for Plasma Glucose Levels
Description: The mean proportional times were evaluated for the following Plasma Glucose Levels: >180 mg/dL, >250 mg/dL, <54 mg/dL, and <70 The mean proportional times evaluated for each Plasma Glucose Level were during the following post-study drug injection periods: 0 to 90 minutes, 0 to 180 minutes, 0 to 360 minutes
Time Frame: Up to 360 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants 0 to 90, 0 to 180, and 0 to 360 minutes after study drug administration with any evaluable plasma glucose concentration data. (While the number of participants noted for each datapoint had evaluable plasma glucose concentration data, not all of the participants had values in the range of plasma glucose concentration required for the analysis of the proportion of time with glucose concentrations in the specified range.)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 17
percentage of time
  >180 mg/dL: 0 to 90 minutes: number analyzed (Participants) | 6 | 3 | 12
  >180 mg/dL: 0 to 90 minutes | 5.6 (13.61) | 0.0 (0.00) | 17.6 (16.72)
  >180 mg/dL: 0 to 180 minutes: number analyzed (Participants) | 14 | 16 | 14
  >180 mg/dL: 0 to 180 minutes | 33.3 (19.61) | 31.3 (13.44) | 58.7 (14.57)
  >180 mg/dL: 0 to 360 minutes: number analyzed (Participants) | 18 | 17 | 14
  >180 mg/dL: 0 to 360 minutes | 45.8 (24.79) | 45.1 (23.21) | 50.8 (18.25)
  >250 mg/dL: 0 to 90 minutes: number analyzed (Participants) | 0 | 0 | 0
  >250 mg/dL: 0 to 180 minutes: number analyzed (Participants) | 11 | 13 | 12
  >250 mg/dL: 0 to 180 minutes | 19.7 (17.98) | 18.0 (15.90) | 40.3 (15.01)
  >250 mg/dL: 0 to 360 minutes: number analyzed (Participants) | 16 | 14 | 12
  >250 mg/dL: 0 to 360 minutes | 27.1 (21.41) | 28.6 (19.81) | 33.3 (16.67)
  <54 mg/dL: 0 to 90 minutes: number analyzed (Participants) | 3 | 4 | 2
  <54 mg/dL: 0 to 90 minutes | 14.8 (16.97) | 19.4 (24.64) | 0 (0)
  <54 mg/dL: 0 to 180 minutes: number analyzed (Participants) | 3 | 4 | 3
  <54 mg/dL: 0 to 180 minutes | 7.4 (8.49) | 9.7 (12.32) | 0 (0)
  <54 mg/dL: 0 to 360 minutes: number analyzed (Participants) | 3 | 4 | 4
  <54 mg/dL: 0 to 360 minutes | 3.7 (4.25) | 43.1 (49.72) | 52.1 (40.15)
  <70 mg/dL: 0 to 90 minutes: number analyzed (Participants) | 5 | 7 | 4
  <70 mg/dL: 0 to 90 minutes | 46.7 (26.53) | 41.3 (25.43) | 19.4 (5.56)
  <70 mg/dL: 0 to 180 minutes: number analyzed (Participants) | 5 | 7 | 5
  <70 mg/dL: 0 to 180 minutes | 30.0 (23.76) | 20.6 (12.72) | 22.2 (34.47)
  <70 mg/dL: 0 to 360 minutes: number analyzed (Participants) | 5 | 8 | 6
  <70 mg/dL: 0 to 360 minutes | 15.0 (11.88) | 28.1 (39.88) | 52.3 (42.33)
Statistical Analysis 1: Comparison: PRAM9 vs Regular Insulin; Plasma Glucose Levels: >180 mg/dL: 0 to 90 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: Means are not equal across the treatment groups; p = 0.041, ANOVA; LS Mean Difference = -21.29, 95% CI 2-sided [-41.23 to -1.36]
Statistical Analysis 2: Comparison: PRAM9 vs Regular Insulin + Pramlintide; Plasma Glucose Levels: >180 mg/dL: 0 to 90 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: Means are not equal across the treatment groups; p = 0.453, ANOVA; LS Mean Difference = -7.45, 95% CI 2-sided [-31.43 to 16.54]
Statistical Analysis 3: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; Plasma Glucose Levels: >180 mg/dL: 0 to 90 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: means are not equal across the treatment groups; p = 0.161, ANOVA; LS Mean Difference = 13.85, 95% CI 2-sided [-8.46 to 36.15]
Statistical Analysis 4: Comparison: PRAM9 vs Regular Insulin; Plasma Glucose >180 mg/dL: 0 to 180 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: means are not equal across the treatment groups; p < 0.001, ANOVA; LS Mean Difference = -23.93, 95% CI 2-sided [-35.37 to -12.48]
Statistical Analysis 5: Comparison: PRAM9 vs Regular Insulin + Pramlintide; Plasma Glucose >180 mg/dL: 0 to 180 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: means are not equal across the treatment groups; p = 0.564, ANOVA; LS Mean Difference = 3.10, 95% CI 2-sided [-7.80 to 14.00]
Statistical Analysis 6: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; Plasma Glucose >180 mg/dL: 0 to 180 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: means are not equal across the treatment groups; p < 0.001, ANOVA; LS Mean Difference = 27.03, 95% CI 2-sided [15.96 to 38.09]
Statistical Analysis 7: Comparison: PRAM9 vs Regular Insulin; Plasma Glucose >180 mg/dL: 0 to 360 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: means are not equal across the treatment groups; p = 0.813, ANOVA; LS Mean Difference = -1.74, 95% CI 2-sided [-16.70 to 13.22]
Statistical Analysis 8: Comparison: PRAM9 vs Regular Insulin + Pramlintide; Plasma Glucose >180 mg/dL: 0 to 360 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: means are not equal across the treatment groups; p = 0.730, ANOVA; LS Mean Difference = 2.35, 95% CI 2-sided [-11.47 to 16.17]
Statistical Analysis 9: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; Plasma Glucose >180 mg/dL: 0 to 360 minutes; Test type: Equivalence — H0: Means are equal between treatment groups. Ha: means are not equal across the treatment groups; p = 0.582, ANOVA; LS Mean Difference = 4.09, 95% CI 2-sided [-10.97 to 19.15]

3. Secondary Outcome: Mean Proportional Time After Glucose Challenge for Plasma Glucose Levels Between 126 to 180 mg/dL
Description: The mean proportional times to plasma glucose levels between 126 to 180 mg/dL following a glucose challenge administered 30 minutes post study drug administration.
Time Frame: During 40 to 180 minutes post-injection of study drug
Population: The number of participants analyzed were the number of participants 0 to 90, 0 to 180, and 0 to 360 minutes after study drug administration with any evaluable plasma glucose concentration data. (While the number of participants noted for each data point had evaluable plasma glucose concentration data, not all of the participants had values in the range of plasma glucose concentration required for the analysis of the proportion of time with glucose concentrations in the specified range.)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 15 | 12 | 16
percentage of time | 11.0 (11.41) | 10.7 (19.38) | 9.8 (11.92)

4. Secondary Outcome: Area Under the Concentration (AUC) Curve for Plasma Glucose
Description: AUC0-t (mg/dL*minutes) for plasma glucose X mg/dL, in which X = (>180 mg/dL, >250 mg/dL) and t = 90, 180, and 360 minutes
Time Frame: Up to 360 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants after study drug administration with evaluable glucose measurements.
  (The time period of 0 to 90 minutes after study drug administration with glucose >250 mg/dL was not quantifiable.)
Measure: Mean (Standard Deviation); unit: min*mg/dL
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 17
min*mg/dL
  AUC 0-90: >180 mg/dL: number analyzed (Participants) | 6 | 3 | 12
  AUC 0-90: >180 mg/dL | 475.0 (1163.51) | 0 (0) | 1108.3 (1193.57)
  AUC 0-180: >180 mg/dL: number analyzed (Participants) | 14 | 16 | 14
  AUC 0-180: >180 mg/dL | 5019.6 (4276.53) | 4591.9 (3095.53) | 13317.5 (5262.42)
  AUC 0-360: >180 mg/dL: number analyzed (Participants) | 18 | 17 | 14
  AUC 0-360: >180 mg/dL | 16255.8 (13128.46) | 16101.2 (11859.68) | 22334.6 (13794.26)
  AUC 0-180: >250 mg/dL: number analyzed (Participants) | 11 | 13 | 12
  AUC 0-180: >250 mg/dL | 1592.7 (1813.87) | 1455.0 (1783.26) | 6302.5 (3495.22)
  AUC 0-360: >250 mg/dL: number analyzed (Participants) | 16 | 14 | 12
  AUC 0-360: >250 mg/dL | 6506.3 (8153.00) | 6847.5 (7282.23) | 16572.5 (26676.00)

5. Secondary Outcome: Area Over the Concentration (AOC) Curve for Plasma Glucose
Description: AOC0-t (mg/dL*minutes) for plasma glucose X mg/dL, in which X = <54 mg/dL and <70 mg/dL and t = 90, 180, and 360 minutes
Time Frame: Up to 360 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants after study drug administration with evaluable glucose measurements.
  (There was no data available for the analysis of AOC0-90 for plasma glucose <54 mg/dL.)
Measure: Mean (Standard Deviation); unit: min*mg/dL
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 17
min*mg/dL
  AUC 0-90: <54 mg/dL: number analyzed (Participants) | 3 | 4 | 2
  AUC 0-90: <54 mg/dL | 658.3 (753.40) | 677.5 (890.36) | 0.0 (0.00)
  AOC 0-180: <54 mg/dL: number analyzed (Participants) | 3 | 4 | 3
  AOC 0-180: <54 mg/dL | 658.3 (753.40) | 677.5 (890.36) | 0 (0)
  AOC 0-360: <54 mg/dL: number analyzed (Participants) | 3 | 4 | 4
  AOC 0-360: <54 mg/dL | 658.3 (753.40) | 3545.0 (6603.37) | 7531.3 (5681.44)
  AOC 0-90: <70 mg/dL: number analyzed (Participants) | 5 | 7 | 4
  AOC 0-90: <70 mg/dL | 2565.0 (1665.80) | 2086.4 (1355.66) | 1010.0 (337.27)
  AOC 0-180: <70 mg/dL: number analyzed (Participants) | 5 | 7 | 5
  AOC 0-180: <70 mg/dL | 3243.0 (2611.35) | 2086.4 (1355.66) | 1874.0 (2587.66)
  AOC 0-360: <70 mg/dL: number analyzed (Participants) | 5 | 8 | 6
  AOC 0-360: <70 mg/dL | 3243.0 (2611.35) | 3797.5 (6070.52) | 8242.5 (6016.84)

6. Secondary Outcome: Plasma Glucose Cmax
Description: The maximum measured glucose concentrations over the time span.
Time Frame: Up to 360 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants after study drug administration with evaluable glucose measurements.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 17
mg/dL | 301.4 (66.72) | 303.3 (73.37) | 339.9 (162.73)

7. Secondary Outcome: Plasma Glucose Tmax
Description: The time to maximum measured glucose concentrations.
Time Frame: Up to 360 minutes following administration of study drug
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 17
minutes | 251.7 (83.68) | 208.3 (47.68) | 150.0 (49.75)

8. Secondary Outcome: Pramlintide Cmax
Description: The maximum measured pramlintide concentrations (arithmetic mean).
Time Frame: Up to 360 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants after study drug administration with evaluable pramlintide measurements.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 0
pg/mL | 99.22 (41.403) | 278.37 (148.512) |
Statistical Analysis 1: Comparison: PRAM9 vs Regular Insulin + Pramlintide; The statistical model was an analysis of variance (ANOVA) on the ln-transformed data with sequence, period, and treatment as fixed effect and subject nested within sequence as a random effect; Test type: Equivalence — Bioequivalence would require 90% confidence intervals of the geometric mean ratio to be contained within the 80-125% range. H0: Means are equal between treatment groups. Ha: Means are not equal across the treatment groups; p < 0.0001, ANOVA — Results of the statistical evaluation of ANOVA (alpha=0.05) for the hypothesis of equal treatment effects; Ratio of geometric least-squares means = 37.04, 90% CI 2-sided [31.36 to 43.75] — Ratio calculated as PRAM geometric least-squares mean divided by the Regular Insulin + Pramlintide geometric least-squares mean, expressed as a percentage. Confidence interval on the ratio, expressed as a percentage

9. Secondary Outcome: Pramlintide Tmax
Description: The time to maximum measured pramlintide concentrations.
Time Frame: Up to 360 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants after study drug administration with evaluable pramlintide concentrations.
Measure: Median (Full Range); unit: minutes
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 0
minutes | 40.5 [21 to 150] | 10.0 [10 to 24] |
Statistical Analysis 1: Comparison: PRAM9 vs Regular Insulin + Pramlintide; The statistical model was an analysis of variance (ANOVA) with sequence, period, and treatment as fixed effect and subject nested within sequence as a random effect; Test type: Other; p < 0.0001, ANOVA — Results of the statistical evaluation of ANOVA (alpha = 0.05) for the hypothesis of equal treatment effects; Ratio of least-square means = 435.96 — Ratio calculated as PRAM least-squares mean divided by the Regular Insulin + Pramlintide least-squares mean, expressed as a percentage

10. Secondary Outcome: Pramlintide Area Under the Concentration (AUC) Curve
Description: The pramlintide area under the concentration time curve after study drug administration (arithmetic mean).
Time Frame: Up to 360 minutes following administration of study drug
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: min*pg/mL
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 0
min*pg/mL
  AUC 0-90 | 5752.239 (2964.0340) | 10317.775 (6782.4249) |
  AUC 0-180 | 9021.278 (4669.0851) | 11079.075 (7836.2702) |
  AUC 0-360 | 9491.208 (4974.9490) | 11132.408 (7948.9301) |
Statistical Analysis 1: Comparison: PRAM9 vs Regular Insulin + Pramlintide; AUC 0 to 90 The statistical model was an analysis of variance (ANOVA) on the ln-transformed data with sequence, period, and treatment as fixed effect and subject nested within sequence as a random effect; Test type: Equivalence — Bioequivalence would require the 90% confidence intervals of the geometric mean ratio to be contained within the 80 - 125% range. H0: Means are equal between treatment groups. Ha: Means are not equal across the treatment groups; p = 0.0075, ANOVA — Results of the statistical evaluation of ANOVA (alpha=0.05) for the hypothesis of equal treatment effects; Ratio of geometric least-squares means = 60.44, 90% CI 2-sided [45.41 to 80.43] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: PRAM9 vs Regular Insulin + Pramlintide; AUC 0 to 180 The statistical model was an analysis of variance (ANOVA) on the ln-transformed data with sequence, period, and treatment as fixed effect and subject nested within sequence as a random effect; Test type: Equivalence — Bioequivalence would require 90% confidence intervals of the geometric mean ratio to be contained within the 80 - 125% range. H0: Means are equal between treatment groups. Ha: Means are not equal across the treatment groups; p = 0.6773, ANOVA — Results of the statistical evaluation of ANOVA (alpha=0.05) for the hypothesis of equal treatment effects; Based on Least-Squares geometric means for ln-transformed data; Ratio of geometric least-squares means = 93.32, 90% CI 2-sided [70.14 to 124.16] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: PRAM9 vs Regular Insulin + Pramlintide; AUC 0 to 360 The statistical model was an analysis of variance (ANOVA) on the ln-transformed data with sequence, period, and treatment as fixed effect and subject nested within sequence as a random effect; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.8768, ANOVA — Results of the statistical evaluation of ANOVA (alpha=0.05) for the hypothesis of equal treatment effects; Ratio of geometric least-squares means = 97.43, 90% CI 2-sided [72.94 to 130.14] — [estimate comment as in outcome 8, analysis 1]

11. Secondary Outcome: Insulin Cmax
Description: The maximum measured insulin concentrations (arithmetic mean)
Time Frame: Up to 360 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants after study drug administration with evaluable insulin measurements.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 17
pg/mL | 724.97 (345.106) | 912.09 (393.686) | 1198.70 (439.528)
Statistical Analysis 1: Comparison: PRAM9 vs Regular Insulin; The statistical model was ana analysis of variance (ANOVA) on the ln-transformed data with sequence, period, and treatment as fixed effect and subject nested within sequence as a random effect; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p < 0.0001, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 53.83, 90% CI 2-sided [44.51 to 65.11] — Ratio calculated as PRAM geometric least-squares mean divided by the Regular Insulin geometric least-squares mean, expressed as a percentage. Confidence interval on the ratio, expressed as a percentage
Statistical Analysis 2: Comparison: PRAM9 vs Regular Insulin + Pramlintide; [analysis description as in outcome 8, analysis 1]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.0192, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 73.16, 90% CI 2-sided [61.06 to 87.67] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; [analysis description as in outcome 8, analysis 1]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.0244, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 135.91, 90% CI 2-sided [113.10 to 163.31] — Ratio calculated as Regular Insulin geometric least-squares mean divided by the Regular Insulin + Pramlintide geometric least-squares mean, expressed as a percentage. Confidence interval on the ratio, expressed as a percentage

12. Secondary Outcome: Insulin Tmax
Description: The time to maximum measured insulin concentrations.
Time Frame: Up to 360 minutes following administration of study drug
Population: The number of participants analyzed were the number of participants after study drug administration with evaluable insulin concentrations.
Measure: Median (Full Range); unit: minutes
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 17
minutes | 120.0 [0 to 241] | 90.5 [40 to 300] | 121.0 [30 to 360]
Statistical Analysis 1: Comparison: PRAM9 vs Regular Insulin; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.2541, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of least-square means = 73.53 — Ratio calculated as PRAM least-squares mean divided by the Regular Insulin least-squares mean, expressed as a percentage
Statistical Analysis 2: Comparison: PRAM9 vs Regular Insulin + Pramlintide; [analysis description as in outcome 9, analysis 1]; Test type: Other; p > 0.9999, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of least-squares means = 103.89 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.1747, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of least-square means = 141.29 — Ratio calculated as Regular Insulin least-squares mean divided by the Regular Insulin + Pramlintide least-squares mean, expressed as a percentage

13. Secondary Outcome: Insulin Area Under the Concentration (AUC) Curve
Description: The insulin area under the concentration time curve after study drug administration.
Time Frame: Up to 360 minutes following administration of study drug
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: min*pg/mL
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
Number analyzed (Participants) | 18 | 18 | 17
min*pg/mL
  AUC 0-90 | 4332.201 (27662.1733) | 52936.566 (25400.6054) | 59727.578 (26405.0845)
  AUC 0-180 | 90807.346 (45238.6643) | 114109.946 (49208.9630) | 143606.541 (54329.1923)
  AUC 0-360: number analyzed (Participants) | 18 | 17 | 17
  AUC 0-360 | 150580.775 (73403.0839) | 182852.584 (100930.8761) | 269913.163 (100898.6768)
Statistical Analysis 1: Comparison: PRAM9 vs Regular Insulin; [analysis description as in outcome 10, analysis 1]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p < 0.0001, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 53.16, 90% CI 2-sided [43.59 to 64.83] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: PRAM9 vs Regular Insulin + Pramlintide; [analysis description as in outcome 10, analysis 1]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.0018, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 65.24, 90% CI 2-sided [54.02 to 78.80] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; [analysis description as in outcome 10, analysis 1]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.2391, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 122.73, 90% CI 2-sided [101.33 to 148.66] — [estimate comment as in outcome 11, analysis 3]
Statistical Analysis 4: Comparison: PRAM9 vs Regular Insulin; [analysis description as in outcome 10, analysis 2]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p < 0.0001, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 54.20, 90% CI 2-sided [47.58 to 61.73] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: PRAM9 vs Regular Insulin + Pramlintide; [analysis description as in outcome 10, analysis 2]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.0002, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 71.29, 90% CI 2-sided [62.99 to 80.69] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; [analysis description as in outcome 10, analysis 2]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.0026, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 131.55, 90% CI 2-sided [116.01 to 149.17] — [estimate comment as in outcome 11, analysis 3]
Statistical Analysis 7: Comparison: PRAM9 vs Regular Insulin; [analysis description as in outcome 10, analysis 3]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p < 0.0001, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 51.34, 90% CI 2-sided [46.74 to 56.39] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: PRAM9 vs Regular Insulin + Pramlintide; [analysis description as in outcome 10, analysis 3]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.0003, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 78.24, 90% CI 2-sided [71.39 to 85.76] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 9: Comparison: Regular Insulin + Pramlintide vs Regular Insulin; [analysis description as in outcome 10, analysis 3]; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p < 0.0001, ANOVA — Bonferroni-adjusted p-value to maintain the overall Type 1 error rate at 0.05; Ratio of geometric least-squares means = 152.41, 90% CI 2-sided [138.91 to 167.22] — [estimate comment as in outcome 11, analysis 3]

ADVERSE EVENTS:
Time Frame: AEs were collected from time of ICF signature to up to the follow-up visit (7 to 11 days of last dose of study drug).
Description: A TEAE with onset on or after the first dose of study drug, any preexisting AE worsened in severity on or after first dose of study drug.
  Assignment of a TEAE to a specific treatment group:
  * treatment received immediately before onset (including Washout Period)
  * If severity increased in a later period, TEAE at increased severity assigned to the treatment received immediately before the increase
  TEAEs missing relationship were assumed to be related to study drug for analysis purposes
Arm/Group | PRAM9 | Regular Insulin + Pramlintide | Regular Insulin
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 10/18 | 9/18 | 10/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRAM9 (N=18) | Regular Insulin + Pramlintide (N=18) | Regular Insulin (N=17)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) — includes administration site conditions
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) — includes administration site conditions
Injection site discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) — includes administration site conditions
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) — includes administration site conditions
Vessel puncture site thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) — includes administration site conditions
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (9) | 8 (13) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT04074317/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04074317/SAP_001.pdf